CLINICAL TRIAL: NCT06793436
Title: Serratus Anterior Plan Block (SAP) and Pectoralis Blocks (PECS I-II) Application After Open Heart Surgery
Brief Title: Serratus Anterior Plan Block (SAP) and Pectoralis Blocks (PECS I-II) After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 17/05/2023
Record Dates: First submitted 2023-05-17; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: prospective randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and surgeons will be unaware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): The patient who has undergone coronary bypass surgery will be taken to the cardiovascular intensive care unit after the surgical procedure. Necessary preparations will be made to make an SAP block. The needle will be advanced superficially or deep to the serratus anterior muscle and 30 mL of local anesthetic (bupivacaine) will be administered to the fascial plane.
  Interventions: Procedure: chest wall blocks
- Group P (Active Comparator): PECS II block is a combination of PECS I and subpectoral local anesthetic injection targeting the lateral cutaneous branches of the intercostal nerves, long thoracic and thoracodorsal nerves. 15mL or local anesthetic (bupivacaine) will be injected into this area (for 15ml PECS I, 30ml total local anesthetic for 15ml PECS II)
  Interventions: Procedure: chest wall blocks

INTERVENTIONS:
Procedure: chest wall blocks — The effects of anterior chest wall blocks (PECS and SAP will be used in this study) performed for postoperative analgesia on pain scores (to be checked with VAS), opioid consumption, length of hospital stay, mobilization time, side effects and complications in the postoperative period will be examined.
  Other Names: postoperative effects

SUMMARY:
It was aimed to examine the effects of anterior chest wall blocks (PECS and SAP will be used in this study) performed for postoperative analgesia on pain scores (to be checked with VAS), opioid consumption, length of hospital stay, duration of mobilization, side effects and complications in the postoperative period.

DETAILED DESCRIPTION:
Patients who were taken in accordance with the inclusion criteria and signed the consent form will be randomly divided into 2 groups. Randomization: Patients will be randomly divided into 2 groups using the closed envelope method:

Group S (Those who will have serratus anterior plane block): The patient who has undergone coronary bypass surgery will be taken to the cardiovascular intensive care unit after the surgical procedure. Necessary preparations will be made to make an SAP block. After ensuring the hygiene of the anterior chest wall, it is advanced with an 8 cm long peripheral block needle under ultrasound guidance. SAP block is a local anesthetic injection procedure applied superficially or deeply to the serratus anterior muscle and specifically targeting the lateral cutaneous and muscular branches of the intercostal nerves. The long thoracic nerve and the thoracodorsal nerve are located in the fascial plane on the surface of the serratus anterior muscle and can be blocked. The serratus anterior block can be performed anywhere between the anterior and posterior axillary lines and the 2nd and 7th ribs. It is performed with the patient in the supine position with the ipsilateral arm abducted 90 degrees or in the lateral decubitus position with the operative side up, while the same side arm is flexed and extended forward. The SAP block will be performed at the level of the 4th rib. The injection site will be found by placing the ultrasound probe under the clavicle in a parasagittal manner and counting from the second rib. By moving the probe laterally towards the mid or posterior axillary line, the serratus anterior muscle will be seen as a layer of muscle over the anechoic shadow of the rib. It extends over the latissimus dorsi serratus anterior muscle and will appear thicker and more prominent in the posterior axillary line. The needle will be advanced superficially or deep to the serratus anterior muscle and 30 mL of local anesthetic (bupivacaine) will be administered to the fascial plane.

Group P (PECS I-II): The patient who has undergone coronary bypass surgery will be taken to the postoperative intensive care unit. Preparation for the PECS block will be made, and after the anterior chest wall hygiene is ensured, an 8 cm long peripheral block needle will be advanced under ultrasound guidance. PECS II block is a combination of PECS I and subpectoral local anesthetic injection targeting the lateral cutaneous branches of the intercostal nerves, long thoracic and thoracodorsal nerves. To perform the PECS I block, the ultrasound probe is placed in the midclavicular line and in the parasagittal plane, and the pectoralis major-minor, axillary vessels and pleura are visualized. After identifying the second and third ribs by sliding the ultrasound probe caudally, the lower end will be rotated towards the axilla to make the probe parallel to the delta pectoral groove. Combined with the in-plane technique, this rotation provides better extension to the intercostobrachial nerve. The tip of the needle will be placed in the interpectoral fascial plane (between pectoralis major and minor) and 15mL of local anesthetic (bupivacaine) will be injected. To perform the PECS II block, in addition to the PECS I block, the needle is advanced from the interpectoral fascial plane to the fascial plane between the pectoralis minor and the serratus anterior. 15mL or local anesthetic (bupivacaine) will be injected into this area (for 15ml PECS I, a total of 30ml local anesthetic for 15ml PECS II). An investigator not associated with the study will perform randomization using a computer generated randomization table. The detection ratio will be 1:1 and sealed opaque envelopes will be used to hide allocations. Outcome assessors and surgeons will be unaware of group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study,
* 20-65 years old
* ASA I-II-III
* Open heart surgery

Exclusion Criteria:

* Refusal to participate in the study
* 20 years old, over 65 years old
* Pregnancy
* Presence of bleeding diathesis
* Liver or kidney failure
* Receiving effective treatment on immunity
* Immune suppressed Those with BMI ≥30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 0,3,6,12. hour Visual analogue scale values
  It will be evaluated with the Visual analogue scale.

SECONDARY OUTCOMES:
side effects and complications | 0,3,6,12. hour
  Side effects and complications after the blocks will be evaluated.
opioid consumption | 0,3,6,12 hours
  The amount of opioid required for analgesic purposes will be monitored after surgery.
number of days in hospital | 1 day
  Length of stay in the intensive care unit after surgery
mobilization time | 1day
  First time mobilized after surgery

CONTACTS AND LOCATIONS:
Overall Officials: School of Mdicine Department of Anesthesiology and Reanimation, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University Faculty of Medicine Department of anesthesiology and reanimation, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' personal information will not be shared.